CLINICAL TRIAL: NCT01588379
Title: Effects of an Afro-centric Dance Program for African-American Daughters and Mothers
Brief Title: Mothers and Girls Dancing Together Trial
Acronym: MAGNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Sofiya Alhassan, Assistant Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0804
Record Dates: First submitted 2012-04-25; First posted 2012-05-01 (Estimated); Last update posted 2023-06-08 (Actual); Status verified 2016-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Girls and mothers dance together (Experimental): African-American girls AND their mom's will participate in the Afro-centric dance program together and also receive weekly newsletter that focuses on health related issues.
  Interventions: Behavioral: Girls and mothers Afro-centric dance program
- Girls, alone (Experimental): African-American girls will participate in the Afro-centric dance program alone. Girls and mom's will receive weekly newsletter that focuses on health related issues
  Interventions: Behavioral: Girls, alone
- No dancing (Active Comparator): African-American girls and their mom's will only receive weekly newsletter that focuses on health related issues.
  Interventions: Other: Newsletter

INTERVENTIONS:
Behavioral: Girls and mothers Afro-centric dance program — African-American girls and their mom's will participate in an after school Afro-centric dance program for 3 days/week for 12 weeks. Both girls and the mothers will also receive weekly newsletter containing various health information.
  Other Names: Girls and mothers, together
  Arms: Girls and mothers dance together
Behavioral: Girls, alone — African-American girls (without their mom's) will participate in an after school Afro-centric dance program for 3 days/week for 12 weeks. Both girls and the mothers will also receive weekly newsletter containing various health information.
  Arms: Girls, alone
Other: Newsletter — Both girls and the mothers will receive weekly newsletter containing various health information.
  Other Names: Control
  Arms: No dancing

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of a 12-week afterschool afro-centric dance physical activity program for daughters and mothers on the physical activity level of African-American girls.

DETAILED DESCRIPTION:
Like African-American women, African-American girls suffer disproportionately from obesity and Type 2 diabetes mellitus. One factor strongly associated with the development of obesity and Type 2 diabetes mellitus disparities in children is low physical activity levels. Low physical activity is more prevalent in African-American girls, pointing to the critical need for effective physical activity interventions. For a physical activity intervention message to be effective among African-American girls, the program must be enjoyable and tailored to African-American girls and women. One possibility for an appropriate physical activity intervention is afro-centric dance, which has strong cultural and historical significance in the African-American community. This form of physical activity may provide girls with sustained bouts of moderate-to-vigorous physical activity. There appears to be a strong positive correlation between parental and children physical activity levels. In the African-American culture, maternal health behaviors in particular have a strong influence on children's health behaviors. Currently, there are no studies that examine the effects of a daughter-mother Afro-centric dance program on the physical activity levels of African-American girls. Therefore, the purpose of this study will be to examine the feasibility and efficacy of a 12-week physical activity intervention consisting of afro-centric dance and its ability to affect the physical activity levels of African-American girls. If investigators identify afro-centric dance as a sustainable form of physical activity for African-American daughters and mothers, investigators can use this intervention to significantly reduce obesity and Type 2 diabetes mellitus in these groups.

ELIGIBILITY:
Inclusion Criteria for Girls:

* 7 -10 yrs old on the date of randomization
* Defined as African-American if her parent/guardian identifies her as such
* No inclusion criteria will be used for mothers

Exclusion Criteria:

* Unable to wear the activity monitor
* Unable to participate in physical activity, require oxygen supplementation for exertion, have a developmental or physical disability preventing participation, cannot increase their physical activity for any reason, uncorrected structural heart disease)
* If girl and/or mother is unable to read, understand, or complete the informed consent or surveys in English.
* Musculoskeletal injuries or disorders that would prevent participation
* Taking diabetes (type 1 or 2), renal diseases, eating disorder, pregnancy medication
* Take medications affecting growth (e.g., insulin, oral hypoglycemic, thyroid hormone)

Ages: 7 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity level at 12-weeks | Baseline, 6-weeks and 12-weeks after study initiation

SECONDARY OUTCOMES:
Changes in body mass index, fasting insulin, and psychosocial | Baseline and 12-weeks after the initiation of the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Sofiya Alhassan, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- Organizations, Churches, and Elementary Schools, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Alhassan S, Nwaokelemeh O, Greever CJ, Burkart S, Ahmadi M, St Laurent CW, Barr-Anderson DJ. Effect of a culturally-tailored mother-daughter physical activity intervention on pre-adolescent African-American girls' physical activity levels. Prev Med Rep. 2018 May 9;11:7-14. doi: 10.1016/j.pmedr.2018.05.009. eCollection 2018 Sep. PMID 30065909